CLINICAL TRIAL: NCT06523205
Title: Evaluation of the Relationships Between Salivary Tenascin C ,IL-4, IL-6, and IL-1β Levels, Smoking and Periodontal Status
Brief Title: Relationships Between Tenascin C, Smoking and Periodontal Status
Status: Not yet recruiting | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Osman Babayigit, Assistant Professor, Necmettin Erbakan University
Other Study IDs: tenascincsmokeperiodontitis
Record Dates: First submitted 2024-07-12; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Periodontitis; Smoking; Periodontal Diseases
Keywords: periodontitis; cytokines; saliva
MeSH Terms: conditions — Periodontitis; Smoking; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- non-smoking - periodontally healthy: participants who reported never smoking and periodontal healthy.
  Interventions: Diagnostic Test: Clinical Measurements and Saliva Sample Collection
- smoking - periodontally healthy: participants who reported smoking >10 cigarettes per day and periodontal healthy.
  Interventions: Diagnostic Test: Clinical Measurements and Saliva Sample Collection
- non-smoking - periodontitis: participants who reported never smoking, with clinical attachment loss ≥3 mm in >30% of sites, with probing depth ≥5 mm in at least six teeth, and with radiographic bone loss extending to or beyond the middle third of the root in the coronal third will be included.
  Interventions: Diagnostic Test: Clinical Measurements and Saliva Sample Collection
- smoking - periodontitis: participants who reported smoking >10 cigarettes per day for >5 years with clinical attachment loss ≥3 mm in >30% of sites, with probing depth ≥5 mm in at least six teeth, and with radiographic bone loss extending to or beyond the middle third of the root in the coronal third will be included.
  Interventions: Diagnostic Test: Clinical Measurements and Saliva Sample Collection

INTERVENTIONS:
Diagnostic Test: Clinical Measurements and Saliva Sample Collection — Saliva samples will be collected from all patients. Clinical parameters will also be recorded. Plaque index (PI) and gingival index (GI) will be recorded at four sites per tooth. Full-mouth probing depth (PD) and clinical attachment level (CAL) will be detailed per tooth at six sites, and the percentage of bleeding areas will be recorded as present or absent within 20 seconds after probing using a binary scoring system. A calibrated periodontologist will record all clinical parameters using manual probing.
  Following sampling, saliva samples will be stored at -80°C until analysis. Concentrations of Tenascin-C, IL-4, IL-6, and IL-1beta will be analyzed by specific enzyme-linked immunosorbent assay (ELISA) kits in saliva samples.

SUMMARY:
The goal of this observational study is to determine if there is a relationship between different periodontal conditions (gingival healthy, stage 2 grade B, stage 2 grade C, stage 3 grade B, stage 3 grade C) and the levels of tenascin C, IL-1 beta, IL-4, and IL-6 in saliva samples from smokers and non-smokers. The main questions it aims to answer are:

Is there a difference in the levels of tenascin C, IL-1 beta, IL-4, and IL-6 between smokers and non-smokers with different periodontal conditions? Do these biomarkers correlate with the severity and grade of periodontal disease?

Researchers will compare the saliva samples from smokers and non-smokers across the different periodontal conditions to see if there are significant differences in the biomarker levels. Participants will:

Provide saliva samples. Be categorized based on their smoking status and periodontal condition.

ELIGIBILITY:
Inclusion Criteria:

* The periodontitis groups (Non-smoking and smoking) in the study will include systemically healthy patients who are clinically diagnosed with Stage II and III, generalized, Grade B, C periodontitis based on the consensus report of the 2017 World Workshop on Classification of Periodontal and Peri-Implant Diseases and Conditions.
* Agreeing to participate in the study

Exclusion Criteria:

* use of oral contraceptive drugs
* use of antibiotics, immunosuppressants, or drug therapies in the last 6 months before the study;
* history of excessive alcohol use;
* pregnancy or breastfeeding status;
* periodontal treatment during the last 6 months before the study.
* Not agreeing to participate in the study
* Not meeting the inclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is planned to be conducted with 100 individuals aged between 18 and 65 who apply to the Department of Periodontology, Faculty of Dentistry, Necmettin Erbakan University, for various reasons. The eligibility of individuals to be included will be evaluated by Assistant Professor Dr. Osman BABAYIGIT at the Periodontology Clinic of NEU Faculty of Dentistry.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
1.Periodontal clinical parameters (plaque index (PI) and gingival index (GI)) | baseline
  The measurements will be performed using a Williams periodontal probe (Hu-Friedy, Chicago, IL, USA) and will include plaque index (PI) and gingival index (GI) at six sites per tooth (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual and disto-lingual) on each tooth.
  Gingival Index (GI) Unit: Numerical score Plaque Index (PI) Unit: Numerical score
Periodontal clinical parameters (percentage bleeding on probing (BOP)) | baseline
  The measurements will be performed using a Williams periodontal probe (Hu-Friedy, Chicago, IL, USA) and will include percentage bleeding on probing (BOP) at six sites per tooth (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual and disto-lingual) on each tooth.
  Percentage Bleeding on Probing (BOP) Unit: Percentage (%)
Periodontal clinical parameters (Clinical Attachment Level (CAL) and Probing Pocket Depth (PPD)) | baseline
  The measurements will be performed using a Williams periodontal probe (Hu-Friedy, Chicago, IL, USA) and will include probing pocket depth (PPD) and clinical attachment level (CAL) at six sites per tooth (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual and disto-lingual) on each tooth.
  Clinical Attachment Level (CAL) Unit: Millimeters (mm) Probing Pocket Depth (PPD) Unit: Millimeters (mm)
Levels of Tenascin C, IL-1β, IL-4 and IL-6 saliva samples | baseline
  Levels of Tenascin C, IL-1β, IL-4 and IL-6 saliva samples (ng/L)
  Unit: Picograms per milliliter (pg/mL)
  Tenascin C, IL-1β, IL-4 and IL-6 levels will be assayed with commercially available kits using the enzyme-linked immunosorbent assay (ELISA) method.

IPD SHARING:
Plan to Share IPD: Undecided